CLINICAL TRIAL: NCT07342244
Title: Safety and Efficacy of CLL1 CAR-T Followed by Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-D
Record Dates: First submitted 2025-12-16; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: AML; AML (Acute Myeloid Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:Experimental group (Experimental): CLL1 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation
  Interventions: Drug: CLL1 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: CLL1 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation — CLL1 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation

SUMMARY:
This study aims to evaluate whether an innovative combination therapy (CLL1 CAR-T sequential allogeneic hematopoietic stem cell transplantation) is safe, feasible and effective for the treatment of relapsed/refractory acute myeloid leukemia (R/R AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients or their guardians understand and voluntarily sign the informed consent form, and are expected to complete the follow-up examinations and treatments as required by the study protocol.

Age between 18-75 years (inclusive), gender not restricted. Confirmed diagnosis of acute myeloid leukemia (AML), with prior receipt of at least one course of systemic chemotherapy, and efficacy assessment showing relapse/refractory disease.

Flow cytometry of bone marrow examination or immunohistochemistry of tumor pathology at screening confirms positive expression of CLL1 target.

Patients have recovered from the toxicity of previous treatments, i.e., CTCAE toxicity grade < 2 (unless the abnormality is tumor-related or judged by the investigator to be in a stable state with little impact on safety or efficacy).

ECOG performance status score 0-2 and expected survival time > 3 months. Adequate organ function:a) Alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)b) Aspartate aminotransferase (AST) ≤ 3 × ULNc) Total bilirubin ≤ 1.5 × ULNd) Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/mine) Hemoglobin ≥ 60 g/L or maintained at this level after blood transfusionf) Indoor oxygen saturation ≥ 92%g) Left ventricular ejection fraction (LVEF) ≥ 45% Capable of establishing venous access required for apheresis, with no contraindications to leukapheresis.

Exclusion Criteria:

* History of other malignancies within 3 years prior to screening, except for adequately treated cervical carcinoma in situ, papillary thyroid carcinoma, basal cell or squamous cell skin carcinoma, locally treated prostate cancer after radical treatment, and ductal carcinoma in situ after radical treatment.

Diagnosis of Waldenström macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary AL amyloidosis at screening.

Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) with HBV DNA titer in peripheral blood above the lower limit of detection of the research institution; positive for hepatitis C virus (HCV) antibody with positive HCV-RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; cytomegalovirus (CMV) DNA quantitative test above the lower limit of detection of the research institution; positive for Treponema pallidum antibody; Epstein-Barr virus (EBV) DNA quantitative test above the lower limit of detection of the research institution.

History of severe allergic reactions [severe allergic reaction is defined as grade 2 or higher allergic reaction, with any of the following clinical manifestations: airway obstruction (runny nose, cough, wheezing, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory or cardiac arrest] or known hypersensitivity to any active ingredients, excipients of the study drugs (including lymphodepletion regimen), murine products, or heterologous proteins.

History of severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, large myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, myocardial infarction or coronary artery bypass grafting (CABG) within ≤ 6 months prior to screening, history of unexplained syncope not due to vasovagal reaction or dehydration, history of severe non-ischemic cardiomyopathy, refractory hypertension (refractory hypertension is defined as: despite lifestyle modifications, blood pressure remains uncontrolled after >1 month of treatment with ≥3 antihypertensive drugs (including diuretics) at reasonable and tolerable maximum doses, or requires ≥4 antihypertensive drugs to effectively control blood pressure).

Unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases requiring medical treatment.

Previous organ transplantation or planned organ transplantation (except hematopoietic stem cell transplantation).

Previous receipt of CAR-T therapy. History of acute/chronic graft-versus-host disease (GVHD) within 6 months prior to screening, or patients requiring immunosuppressive therapy for GVHD.

Active autoimmune or inflammatory neurological diseases (e.g., Guillain-Barré syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).

Presence of tumor emergencies (e.g., spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) requiring urgent treatment at screening or before infusion.

Uncontrolled bacterial, fungal, viral or other infections requiring antibiotic treatment.

Use of short-acting hematopoietic cytokines affecting blood counts within 1 week prior to planned blood collection for CAR-T manufacturing, or use of long-acting hematopoietic cytokines within 2 weeks prior to screening, and judged by the investigator to have an impact on cell manufacturing.

Receipt of corticosteroids or immunosuppressive drugs within 2 weeks prior to planned blood collection for CAR-T manufacturing at screening, and judged by the investigator to have an impact on cell manufacturing:a) Corticosteroids: Subjects receiving systemic steroid therapy within 2 weeks prior to planned blood collection for CAR-T manufacturing at screening and judged by the investigator to require long-term systemic steroid therapy during treatment (except inhaled or topical use); and subjects receiving systemic steroid therapy within 72 hours before cell infusion (except inhaled or topical use).b) Immunosuppressants: Subjects receiving immunosuppressive therapy within 2 weeks prior to planned blood collection for CAR-T manufacturing at screening.

Major surgical procedures (except diagnostic surgery and biopsy) within 4 weeks prior to lymphodepletion or planned major surgery during the study period, or surgical wounds not fully healed before enrollment.

Vaccination with (attenuated) live viral vaccines within 4 weeks prior to screening.

Presence of severe mental illness. History of alcoholism or drug abuse. Pregnant or lactating women, and female subjects planning pregnancy within 2 years after cell infusion or male subjects whose partners plan pregnancy within 2 years after their cell infusion.

Subjects with contraindications to any study procedures or other medical conditions that may expose them to unacceptable risks, as judged by the investigator and/or according to clinical standards.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1,3,6,12,18,24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China